CLINICAL TRIAL: NCT07256717
Title: Balanced Progressive Intensity Training (BPIT): A Five-Week Multi-Site Clinical Evaluation of Functional Movement, Mobility, and Neuromuscular Adaptation in Healthy Adults (18-65 Years)
Brief Title: BPIT 5-Week Multi-Site Study: Movement Efficiency, Mobility & Neuromuscular Adaptation
Acronym: BPIT_5LINE_369
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MMSx Authority Institute for Movement Mechanics & Biomechanics Research Inc. (Other)
Collaborators: BodyGNTX Fitness Institute (Unknown); GFFI Fitness Academy (Unknown); Indian Institute of Kinesiology and Biomechanics Science (IIKBS) (Unknown); Bureau of Fitness Standards (BFS) (Unknown); Active India Health & Fitness Trust (AIHFT) (Unknown); Body Mechanic Chain of Gyms (Unknown); Shri Mahaveer Ortho Clinic (Unknown); Regain Fitness Zone (Unknown); MMSx Authority Biomechanics Department (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BPIT-MULTI-2025-001; MACREB-BPIT-2025-014 (Other: nstitutional Ethics Committee Approval Number (MMSx Authority / GFFI Ethics Committee))
Record Dates: First submitted 2025-11-18; First posted 2025-12-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Physical Fitness
Keywords: Balanced Progressive Intensity Training; BPIT; 5-Line Principle; Movement Efficiency; Heart Rate Variability; Postural Control; Strength Training; Exercise Intervention; Neuromuscular Adaptation

STUDY DESIGN:
Masking Description: Single-arm prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPIT 5-Line Training Group (Experimental): All participants receive the 5-week Balanced Progressive Intensity Training (BPIT) program using the 5-Line Principle (ground-based → knee-level → standing → head-level → plyometric) under supervised sessions 3-5 times per week.
  Interventions: Behavioral: Balanced Progressive Intensity Training (BPIT) 5-Line Method

INTERVENTIONS:
Behavioral: Balanced Progressive Intensity Training (BPIT) 5-Line Method — 5-week supervised progressive training using the BPIT 5-Line framework developed by Dr. Neeraj Mehta.

SUMMARY:
This prospective, multi-site, single-arm interventional study evaluates the 5-Line Principle of Balanced Progressive Intensity Training (BPIT) over 5 weeks in healthy adults aged 18-65 years. All participants receive supervised BPIT sessions (3-5 per week) progressing through five intensity lines defined by anatomical landmarks and ground reaction force:

Ground-Based (Low) Knee-Level (Low-Moderate) Standing (Moderate) Head-Level (Moderate-High) Plyometric (High-Impact)

The study aims to quantify improvements in functional movement efficiency, joint mobility, postural control, strength adaptation, and heart-rate variability while monitoring safety and individual overload indicators.

DETAILED DESCRIPTION:
Primary Outcome Measures

Change in Functional Movement Screen (FMS) total score from baseline to Week 5 Change in Y-Balance Test reach distance (composite score) Timeframe: Baseline and Week 5

Secondary Outcome Measures

Change in 1-RM or estimated strength (squat, deadlift, overhead press) Change in resting HRV (RMSSD) Change in joint range of motion (goniometry) and postural sway Incidence of training-related discomfort or minor injury Timeframe: Baseline, weekly, and Week 5

Arms/Intervention Experimental: BPIT 5-Line Training Group Intervention: Behavioral: Balanced Progressive Intensity Training (BPIT) 5-Line Method Description: 5-week supervised progressive training using the BPIT 5-Line framework (ground-based → plyometric) Eligibility

Ages Eligible: 18 Years to 65 Years Sexes Eligible: All Accepts Healthy Volunteers: Yes

Inclusion Criteria

Healthy adults with regular exercise history Able to attend 3-5 training sessions/week Signed informed consent

Exclusion Criteria

Recent injury (<3 months) Known cardiovascular, metabolic, or orthopaedic contraindications Pregnancy

Study Locations 13 Locations in India 2 Locations in USA, (Details of the location is uploaded on mmsxauthority.com webiste)

MMSx Authority , USA, GFFI Fitness Academy, New Delhi BodyGNTX USA BFS/AIHFT-approved facilities

Countries of Recruitment India U.S. FDA-regulated? No / No / No Human Subjects Protection Review Board Status Approved (or Submit for review if not yet) Board Name: Institutional Ethics Committee - MMSx Authority / GFFI Approval Number: BPIT-MULTI-2025-001 (or pending) Data Monitoring Committee No

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years Generally healthy with regular physical activity history (at least 1-2 sessions per week for the past 3 months) Able to commit to 3-5 supervised training sessions per week for 5 weeks Willing and able to provide written informed consent Cleared by pre-screening (no acute injury, no contraindications)

Exclusion Criteria:

* Acute musculoskeletal injury within the past 3 months Known cardiovascular, metabolic, or orthopaedic conditions that contraindicate exercise Pregnancy or planning pregnancy Use of medications or supplements that significantly affect muscle recovery or performance (e.g., corticosteroids, anabolic agents) Inability to follow the BPIT protocol or attend required sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Movement Efficiency Score (MES, 0-10) | Baseline (Week 0) and end of study (Week 5)
  Change from baseline in the proprietary Movement Efficiency Score (MES), a validated composite metric of biomechanical function, movement quality, and postural alignment (derived from MMSx Flaw Checklist, visual/video analysis, and functional mapping).

SECONDARY OUTCOMES:
Range of Motion (ROM) | Baseline and Week 5
  Change from baseline in joint range of motion (degrees) measured by goniometry at key sites (shoulder, hip, spine, ankle).
VAS Pain Score | Baseline and Week 5
  Change from baseline in participant-reported pain/discomfort on a 0-10 Visual Analog Scale.
Strength Index | Baseline and Week 5
  Change from baseline in Strength Index calculated as Reps × Load (or estimated 1RM where applicable) for key movements.
Mobility Limitation (%) | Baseline and Week 5
  Change from baseline in self-reported percentage limitation in daily functional tasks due to mobility restrictions.

OTHER OUTCOMES:
Heart Rate Variability (HRV - RMSSD) | Baseline and Week 5
  Change from baseline in resting heart rate variability (RMSSD) as a biomarker of autonomic recovery.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - BodyGNTX Fitness Institute, Columbus, Ohio
  - MMSx Authority Biomechanics Department, Powell, Ohio
  - MMSx AUTHORITY INSTITUTE FOR MOVEMENT MECHANICS & BIOMECHANICS RESEARCH (COORDINATING CENTER), Powell, Ohio
- India (7):
  - Indian Institute of Kinesiology & Biomechanics Science (IIKBS), Burhānpur, Madhya Pradesh
  - Shri Mahaveer Ortho Clinic, Delhi, National Capital Territory of Delhi
  - GFFI Fitness Academy, New Delhi, National Capital Territory of Delhi
  - Active India Health & Fitness Trust (AIHFT), New Delhi, National Capital Territory of Delhi
  - Body Mechanics Gym P Ltd, New Delhi, National Capital Territory of Delhi
  - Regain Fitness Zone, Greater Noida, Uttar Pardesh
  - GFFI Fitness Academy, Agra, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT07256717/Prot_003.pdf
  • Statistical Analysis Plan (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT07256717/SAP_001.pdf
  • Informed Consent Form (2025-11-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT07256717/ICF_002.pdf